CLINICAL TRIAL: NCT00074685
Title: Research Registry for Inherited Disorders of Keratinization
Brief Title: National Registry for Ichthyosis and Related Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: NIAMS-101
Record Dates: First submitted 2003-12-18; First posted 2003-12-19 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2009-04

CONDITIONS: Darier Disease; Hailey-Hailey Disease; Hyperkeratosis, Epidermolytic; Ichthyosis; Ichthyosis, Lamellar; Ichthyosis, X-Linked; Keratoderma
Keywords: Congenital; Epidermal nevus; Erythroderma; Darier; Hailey-Hailey; Harlequin; Ichthyosiform; Ichthyosiform erythroderma; Keratoderma; Keratosis; Pachyonychia; Sjogren-Larsson
MeSH Terms: conditions — Darier Disease; Pemphigus, Benign Familial; Hyperkeratosis, Epidermolytic; Ichthyosis; Ichthyosis, Lamellar; Ichthyosis, X-Linked; Epidermal Nevus; Dermatitis, Exfoliative; Ichthyosiform Erythroderma, Congenital; Keratosis; Nails, Malformed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Histology, DNA from participating enrollees
Oversight: Data Monitoring Committee: No

SUMMARY:
The ichthyoses are a family of genetic skin diseases characterized by dry, thickened, scaling skin. Dermatologists estimate that there are over twenty varieties of ichthyosis, with a wide range of severity and associated symptoms. This registry is designed to identify people in the United States with the ichthyoses and other related disorders and to collect information about their skin ailment and how it has affected them. The database is available for review by approved research applicants. The registry is confidential and provides investigators a way to share information about studies and trials with potential participants while maintaining participants' privacy.

Although the Registry is closed to new enrollment, it is still maintained in order to provide information related to understanding the diagnosis, pathophysiology, and treatment of ichthyoses. Support for studies continues and inquiries from investigators are welcomed.

DETAILED DESCRIPTION:
The purpose of this registry is to support studies aimed at determining the cause of the ichthyoses and treating them more effectively. The Registry offers blinded information about well-characterized groups of individuals with specific diagnoses for study by skin biologists, pharmacologists, and others. The Registry also provides information about research projects to those that have enrolled in the Registry and expressed an interest in participating in studies.

Participants enrolled in the Registry by contacting the registry officials. All participants participated in a phone interview with the study research nurse. Participants were asked about diagnostic testing, treatments, birth history, medical history, degree and type of involvement, current physical condition, and other family members with skin disorders. A quality of life index was embedded in the interview. Participants also indicated whether they would like to be contacted about participating in clinical research. This information was complemented by an enrollment form from the enrollee's caregiver.

Diagnosis was confirmed by specific criteria based on clinical involvement, review of histology, and where appropriate, serum cholesterol sulfate determination or DNA analysis.

ELIGIBILITY:
Note: Accrual into this study has been discontinued as of 03/31/04.

Inclusion Criteria:

* Diagnosis of one of the ichthyoses, erythrokeratodermas, Darier disease, Hailey-Hailey disease, palmar-plantar keratodermas, pachyonychia congenita, extensive epidermal nevi, or related disorder

Exclusion Criteria:

* Ichthyosis Vulgaris

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with one of the following diseases: Erythrokeratoderma, Extensive Epidermal Nevi, Darier disease, Hailey-Hailey disease, Ichthyosis, Palmar-Plantar Keratoderma, or Pachyonychia Congenita
Sampling Method: Non-Probability Sample
Enrollment: 610 (Actual)
Dates: Start 1994-09; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Fleckman, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Fleckman P. Management of the ichthyoses. Skin Therapy Lett. 2003 Sep;8(6):3-7. PMID 14610614
- [Background] Mayes MD, Giannini EH, Pachman LM, Buyon JP, Fleckman P. Connective tissue disease registries. Arthritis Rheum. 1997 Sep;40(9):1556-9. doi: 10.1002/art.1780400903. No abstract available. PMID 9324008
- [Background] Fleckman P: The ichthyosis registry - a resource ready for use. J Invest Dermatol 123(1):x, 2004
- [Result] Richard G, Smith LE, Bailey RA, Itin P, Hohl D, Epstein EH Jr, DiGiovanna JJ, Compton JG, Bale SJ. Mutations in the human connexin gene GJB3 cause erythrokeratodermia variabilis. Nat Genet. 1998 Dec;20(4):366-9. doi: 10.1038/3840. PMID 9843209
- [Result] Zettersten E, Man MQ, Sato J, Denda M, Farrell A, Ghadially R, Williams ML, Feingold KR, Elias PM. Recessive x-linked ichthyosis: role of cholesterol-sulfate accumulation in the barrier abnormality. J Invest Dermatol. 1998 Nov;111(5):784-90. doi: 10.1046/j.1523-1747.1998.00386.x. PMID 9804339
- [Result] Sprecher E, Chavanas S, DiGiovanna JJ, Amin S, Nielsen K, Prendiville JS, Silverman R, Esterly NB, Spraker MK, Guelig E, de Luna ML, Williams ML, Buehler B, Siegfried EC, Van Maldergem L, Pfendner E, Bale SJ, Uitto J, Hovnanian A, Richard G. The spectrum of pathogenic mutations in SPINK5 in 19 families with Netherton syndrome: implications for mutation detection and first case of prenatal diagnosis. J Invest Dermatol. 2001 Aug;117(2):179-87. doi: 10.1046/j.1523-1747.2001.01389.x. PMID 11511292
- [Result] Richard G, Rouan F, Willoughby CE, Brown N, Chung P, Ryynanen M, Jabs EW, Bale SJ, DiGiovanna JJ, Uitto J, Russell L. Missense mutations in GJB2 encoding connexin-26 cause the ectodermal dysplasia keratitis-ichthyosis-deafness syndrome. Am J Hum Genet. 2002 May;70(5):1341-8. doi: 10.1086/339986. Epub 2002 Mar 22. PMID 11912510
- [Result] Richard G, Brown N, Rouan F, Van der Schroeff JG, Bijlsma E, Eichenfield LF, Sybert VP, Greer KE, Hogan P, Campanelli C, Compton JG, Bale SJ, DiGiovanna JJ, Uitto J. Genetic heterogeneity in erythrokeratodermia variabilis: novel mutations in the connexin gene GJB4 (Cx30.3) and genotype-phenotype correlations. J Invest Dermatol. 2003 Apr;120(4):601-9. doi: 10.1046/j.1523-1747.2003.12080.x. PMID 12648223
- [Result] Fowler AJ, Moskowitz DG, Wong A, Cohen SP, Williams ML, Heyman MB. Nutritional status and gastrointestinal structure and function in children with ichthyosis and growth failure. J Pediatr Gastroenterol Nutr. 2004 Feb;38(2):164-9. doi: 10.1097/00005176-200402000-00012. PMID 14734878
- [Result] Moskowitz DG, Fowler AJ, Heyman MB, Cohen SP, Crumrine D, Elias PM, Williams ML. Pathophysiologic basis for growth failure in children with ichthyosis: an evaluation of cutaneous ultrastructure, epidermal permeability barrier function, and energy expenditure. J Pediatr. 2004 Jul;145(1):82-92. doi: 10.1016/j.jpeds.2004.03.052. PMID 15238912
- [Result] Leachman SA, Kaspar RL, Fleckman P, Florell SR, Smith FJ, McLean WH, Lunny DP, Milstone LM, van Steensel MA, Munro CS, O'Toole EA, Celebi JT, Kansky A, Lane EB. Clinical and pathological features of pachyonychia congenita. J Investig Dermatol Symp Proc. 2005 Oct;10(1):3-17. doi: 10.1111/j.1087-0024.2005.10202.x. PMID 16250204
- [Result] Richard G, Ratajcaz P, Amin S, Ilyas H. Netherton Syndrome: Novel and Recurrent Mutations in SPINK5 and implications for screening and diagnosis. J Invest Dermatol 122, 2004.
- [Result] Ross R, DiGiovanna JJ, Capaldi L, Argenyi Z, Fleckman P, Robinson-Bostom L. Histopathologic characterization of epidermolytic hyperkeratosis: a systematic review of histology from the National Registry for Ichthyosis and Related Skin Disorders. J Am Acad Dermatol. 2008 Jul;59(1):86-90. doi: 10.1016/j.jaad.2008.02.031. PMID 18571597
- [Result] Farasat S, Wei MH, Herman M, Liewehr DJ, Steinberg SM, Bale SJ, Fleckman P, Toro JR. Novel transglutaminase-1 mutations and genotype-phenotype investigations of 104 patients with autosomal recessive congenital ichthyosis in the USA. J Med Genet. 2009 Feb;46(2):103-11. doi: 10.1136/jmg.2008.060905. Epub 2008 Oct 23. PMID 18948357
- [Result] Herman ML, Farasat S, Steinbach PJ, Wei MH, Toure O, Fleckman P, Blake P, Bale SJ, Toro JR. Transglutaminase-1 gene mutations in autosomal recessive congenital ichthyosis: summary of mutations (including 23 novel) and modeling of TGase-1. Hum Mutat. 2009 Apr;30(4):537-47. doi: 10.1002/humu.20952. PMID 19241467
- See also: The National Registry for Ichthyosis and Related Disorders — http://www.skinregistry.org
- See also: FIRST - Foundation for Ichthyosis and Related Skin Types — http://www.scalyskin.org